CLINICAL TRIAL: NCT06077201
Title: Home-Based Cardiac Rehabilitation Using a Novel Mobile Health Exercise Regimen Following Transcatheter Heart Valve Interventions
Acronym: HOMERUNHITTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Medical University of South Carolina (Other); University of Pittsburgh (Other); Duke Clinical Research Institute (Other); National Institute on Aging (NIA) (NIH); University of Michigan (Other); The Cleveland Clinic (Other); University of Colorado, Denver (Other); Piedmont Healthcare (Other); Wake Forest University Health Sciences (Other); Morristown Medical Center (Other)
Responsible Party: Principal Investigator, Brian Lindman, Medical Director, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 222231; 5R01AG073633-02 (NIH)
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Valvular Heart Disease
Keywords: cardiac rehabilitation; transcatheter heart valve intervention; cardiology; aortic stenosis; mitral regurgitation; tricuspid regurgitation
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1:1 to 3 groups.
Who Masked: Outcomes Assessor
Masking Description: Study coordinator performing the remote study visits will be blinded to the treatment group allocation until the participant has completed the study visit assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Standard of care course for an individual not participating in center based cardiac rehabilitation. AHA Life's Essential 8 Fact Sheets are provided to promote healthy living.
- HBCR hands-off (Experimental): Home-based cardiac rehabilitation with mobile application + AHA Life's Essential 8 sheets.
  Interventions: Other: HBCR hands-off
- HBCR interactive (Experimental): Home-based cardiac rehabilitation with mobile application and periodic video calls with exercise physiologist + AHA Life's Essential 8 sheets.
  Interventions: Other: HBCR interactive

INTERVENTIONS:
Other: HBCR hands-off — Home-based cardiac rehabilitation intervention facilitated by a custom app to deliver education, counseling on healthy living and modification of risk factors, mindfulness, and physical activity guidance.
  Arms: HBCR hands-off
Other: HBCR interactive — Home-based cardiac rehabilitation intervention facilitated by a custom app to deliver education, counseling on healthy living and modification of risk factors, mindfulness, and physical activity guidance. Additionally, there are periodic video calls with an exercise physiologist.
  Arms: HBCR interactive

SUMMARY:
The vast majority of cardiac rehabilitation eligible individuals do not participate in center based cardiac rehabilitation (CBCR). While steps to encourage participation in CBCR are important, many individuals will still not participate for a variety of reasons. This randomized controlled trial is evaluating a home-based cardiac rehabilitation (HBCR) intervention delivered using a custom app and digital tools in patients undergoing transcatheter heart valve interventions (THVIs). After a brief roll-in period, participants not intending to participate in CBCR are randomized to one of three groups: (1) control, (2) HBCR mobile health intervention with hands-off delivery, and (3) HBCR mobile health intervention with interactive delivery. Participants in the intervention groups (hands-off/interactive delivery) will also be randomized to continue the intervention for 12 weeks or 24 weeks. The intervention targets key health behaviors and includes traditional cardiac rehabilitation components. The study will assess the effect of the intervention on clinical events, physical activity, quality of life, and other outcomes. Those who intend to participate in CBCR will be followed in a registry.

ELIGIBILITY:
Inclusion Criteria:

* Treated with a transcatheter heart valve intervention (e.g., transcatheter aortic valve implantation [in the native valve or valve-in-valve], mitral transcatheter edge-to-edge repair, mitral valve-in-valve) of the aortic, mitral, or tricuspid valve done via transfemoral access

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Not adherent to wearing the ActiGraph activity tracker during the roll-in phase for a minimum of 4 (out of 7) compliant days (worn >10 hours/day)
* Planned participation in center based cardiac rehabilitation (CBCR)
* Transcatheter heart valve intervention done via any route other than a transfemoral approach
* Stroke during or immediately after the transcatheter heart valve intervention prior to randomization
* Placement of a pacemaker within 6 weeks prior to the transcatheter heart valve intervention or after the transcatheter heart valve intervention and prior to randomization
* Those who require a walker or who cannot get out of a chair/bed on their own and walk independently (use of a cane is acceptable)
* Physical or neuropsychiatric limitations that would prevent proficient use of the study tools and successful completion of the physical and quality of life assessments (e.g. blindness, dementia)
* Planned surgery within 6 months after the heart valve intervention
* Planned discharge from hospital to hospice, assisted living, or inpatient rehabilitation facility (discharge to a senior facility permitted as long as they are considered Independent Living)
* Treating provider or site PI indicates that participation in the study would be unsafe
* Participation in any ongoing randomized trial that has not completed follow-up unless the sponsor of the other trial allows enrollment of the participant in this cardiac rehabilitation trial
* Unable to complete the baseline study visit prior to 6 weeks after the transcatheter heart valve intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Probability of the hierarchical clinical event composite | Over the entire available follow-up period for randomized participants (minimum of 6 months, maximum approximately 24-30 months).
  The hierarchical clinical event composite includes (in order of hierarchy): (1) all-cause death; (2) all-cause hospitalization; and (3) skilled nursing facility visits. To examine whether the intervention improves mortality, hospitalization, and SNF rates after THVIs, we will conduct Bayesian Markov longitudinal proportional odds model on weekly outcome measures. The pooled active treatment vs. control group comparison (primary comparison for the trial) will be estimated by contrasting the average of posterior probability that Y≥y of the two active treatment groups (hands-off HBCR and interactive HBCR) to the control group.
Average daily total activity counts | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily total activity counts determined. The primary comparison will be at 12 weeks after randomization.
  Daily total activity counts are determined by a triaxial actigraphy device.

SECONDARY OUTCOMES:
Average daily total activity counts | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily total activity counts determined. The secondary comparisons will be at 24 and 52 weeks after randomization.
  Daily total activity counts are determined by a triaxial actigraphy device.
Average daily active minutes | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily active minutes determined. The comparisons will be at 12, 24 and 52 weeks after randomization.
  Daily active minutes are determined by a triaxial actigraphy device.
Average daily steps | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily steps determined. The comparisons will be at 12, 24 and 52 weeks after randomization.
  Daily steps are determined by a triaxial actigraphy device.
Average daily energy expenditure | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily energy expenditure determined. The comparisons will be at 12, 24 and 52 weeks after randomization.
  Daily energy expenditure is determined by a triaxial actigraphy device.
Average daily moderate to vigorous active minutes | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily moderate to vigorous active mins determined. The comparisons will be at 12, 24 and 52 weeks after randomization.
  Daily moderate to vigorous active minutes are determined by a triaxial actigraphy device.
6 minute walk distance | The comparisons will be at 12, 24 and 52 weeks after randomization.
  The distance walked in 6 minutes.
Chair sit to stand time | The comparisons will be at 12, 24 and 52 weeks after randomization.
  The time taken to complete 5 chair rises.
5 meter gait speed | The comparisons will be at 12, 24 and 52 weeks after randomization.
  The speed of walking 5 meters (meters/second).
All-cause hospitalizations | Over the entire available follow-up period for randomized participants (minimum of 6 months, maximum approximately 24-30 months).
  Hospitalizations for any reason
All-cause death | Over the entire available follow-up period for randomized participants (minimum of 6 months, maximum approximately 24-30 months).
  Death for any cause
Heart-failure specific health status assessed by the KCCQ | The comparisons will be at 12, 24 and 52 weeks after randomization.
  Assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ); (score range 0-100, higher is better health status)
Physical health status assessed by the PROMIS 10 | The comparisons will be at 12, 24 and 52 weeks after randomization.
  Global physical health score from the PROMIS 10 Global Health Short Form questionnaire (raw score range 4-20 with corresponding T score and SE, higher is better)
Mental health status assessed by the PROMIS 10 | The comparisons will be at 12, 24 and 52 weeks after randomization.
  Global mental health score from the PROMIS 10 Global Health Short Form questionnaire (raw score range 4-20 with corresponding T score and SE, higher is better)
Mood disturbance assessed by PHQ9 | The comparisons will be at 12, 24 and 52 weeks after randomization.
  Patient health questionnaire 9 (PHQ9); (score range 1-27, higher score worse)
Patient goals progress score | The comparisons will be at 12, 24 and 52 weeks after randomization.
  A patient goals progress score (-3 to +3) will be determined for 5 domains and the scores combined for a global score from -15 to +15.
Basic mobility by AM-PAC | The comparisons will be at 12, 24 and 52 weeks after randomization.
  Basic mobility will be assessed with the Activity Measure for Post-Acute Care (AM-PAC) Basic Mobility Outpatient Short Form (Low Function); (raw score range 0-39 with corresponding T-score and SE, higher score is better)

CONTACTS AND LOCATIONS:
Overall Officials: Brian R. Lindman, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States